CLINICAL TRIAL: NCT07134569
Title: Motor Function Assessment and VR-based Motor Training in Adults With Autism Spectrum Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202311005RINC
Record Dates: First submitted 2025-02-04; First posted 2025-08-21 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Autism
Keywords: Virtual Reality; motor training
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autism (Experimental)
  Interventions: Behavioral: VR-based motor training
- Typically developing control (No Intervention)

INTERVENTIONS:
Behavioral: VR-based motor training — Six weeks, twice per week.
  Arms: Autism

SUMMARY:
The goal of this clinical trial is to learn if autism affect motor functions, including muscle strength, balance, and motor control? Additionally, understanding the motor functions, cognitive functions, and brain activation in individuals with autism, and verifying whether motor training can effectively improve muscle strength, balance, and motor control. The main questions aim to answer are:

[primary hypothesis or outcome measure 1]? [primary hypothesis or outcome measure 2]? If there is a comparison group: Researchers will compare [arm information] to see if [insert effects].

Participants will [describe the main tasks participants will be asked to do, interventions they'll be given and use bullets if it is more than 2 items].

ELIGIBILITY:
> The ASD Group

Inclusion criteria:

* young adult aged between 18 and 45 years who had a diagnosis of ASD from a licensed mental health or medical professional based on DSM-5.
* was motivated to complete the 6-week VR-based motor function training.
* had a full-scale IQ > 70 on the WAIS-IV.

Exclusion criteria:

* a history of major mental illness (e.g., bipolar affective disorder, schizophrenia, or psychosis), neurological diseases (e.g., stroke, lumbar radiculopathy, or spinal cord injury) that hamper walking function, or neurosurgery.
* visual impairment and/or hearing impairment that would preclude participation in motor assessment or training.

  * The Non-ASD control group

Inclusion criteria:

* young adult aged between 18 and 45 years who do not have a diagnosis of ASD.
* had a full-scale IQ > 70 on the WAIS-IV.

Exclusion criteria:

* a history of major mental illness (e.g., bipolar affective disorder, schizophrenia, or psychosis), neurological diseases (e.g., stroke, lumbar radiculopathy, or spinal cord injury), or neurosurgery that hamper walking function.
* visual impairment and/or hearing impairment that would preclude participation in motor assessment or training.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
The performance of movement operational assessment | 40 minutes
  Participants will take movement operational assessment, which composed of different tests, such as Timed Up and Go Test (TUG), the 10-meter walk test (10MWT) and the 6-minute walk test (6WMT)
The performance of motor coordination control | 1 hour, twice
  the performance recorded with Vicon, an motion capture system, and Single Leg Stance Test

SECONDARY OUTCOMES:
The N-back Task performance | 40 minutes
The performance of Timed Up and Go Test (TUG) | 1 minute, twice
The performance of the 10-meter walk test (10MWT) | 1 minute, twice
The performance of 6-minute walk test (6WMT) | 6 minutes, twice

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan